CLINICAL TRIAL: NCT03217448
Title: The Efficacy and Safety of Dabigatran Etexilate Comparing With Warfarin for the Anticoagulation Treatment of Cerebral Venous Thrombosis :a Pilot Study
Brief Title: The Efficacy and Safety of Dabigatran Etexilate for the Treatment of Cerebral Venous Thrombosis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Ji Xunming, Professor, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DE-CVT
Record Dates: First submitted 2017-07-12; First posted 2017-07-14 (Actual); Last update posted 2017-11-22 (Actual); Status verified 2017-11

CONDITIONS: Cerebral Venous Thrombosis
MeSH Terms: conditions — Intracranial Thrombosis | interventions — Dabigatran; Warfarin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dabigatran etexilate group (Experimental): Subjects in this group will take Dabigatran etexilate for 6 months after randomization
  Interventions: Drug: Dabigatran etexilate
- Warfarin group (Active Comparator): Subjects in this group will take Warfarin for 6 months after randomization
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: Dabigatran etexilate — Subjects should take Dabigatran etexilate 150mg twice a day for 6 months after randomization.
  Arms: Dabigatran etexilate group
Drug: Warfarin — Subjects should take Warfarin for 6 months after randomization and the dose will be changed according to investigator's judgment.
  Arms: Warfarin group

SUMMARY:
This is a single-center, prospective, randomized (1:1), open-label study with two parallel groups. This study is planned to investigate the efficacy and safety of dabigatran etexilate comparing with warfarin for the treatment of cerebral venous thrombosis.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Cerebral Venous thrombosis (CVT), with or without intracranial haemorrhage.
* Patients in the acute or sub-acute phase of CVT.
* Completion of anticoagulation therapy for 5-15 days which has been administered until randomization; anticoagulation must include full-dose low molecular weight heparin or unfractionated heparin.
* Eligibility for treatment with an oral anticoagulant.
* Written informed consent.

Exclusion Criteria:

* Cerebral Venous thrombosis (CVT) associated with central nervous system infection or due to head trauma.
* Thrombosed venous sinuses showed completely recanalized by MRV before randomisation.
* Planned endovascular treatment for CVT or surgical treatment for other diseases.
* Conditions associated with increased risk of bleeding.
* History of symptomatic non-traumatic intracranial haemorrhage with increased risk of recurrence according to investigator's judgment.
* Treatment with an antithrombotic regimen for an indication other than CVT and requiring continuation of that treatment for the original diagnosis.
* Severe renal impairment(CrCL<30mL/min).
* Active liver disease (ALT≥ twice the upper limit of normal).
* Preganancy, nursing or planning to become pregnant during the trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-10-30 (Actual); Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
The incidence of recanalized cerebral veins after 6 months | 0-6 months after randomization
  cerebral venous recanalisation rate after anticoagulation treatment for 6 months.

SECONDARY OUTCOMES:
Number of subjects with venous thrombosis events | 0-6 months after randomization
  Number of subjects with recurrent cerebral venous and dural sinus thrombosis, deep venous thrombosis of any limb, pulmonary embolism or splanchnic vein thrombosis within 6 months.
The change of optic disc edema grade and lumbar puncture pressure after 6 months | 0-6 months after randomization
Number of subjects with major bleeding events | 0-6 months after randomization
  Number of subjects with major bleeding events according to International Society on Thrombosis and Haemostasis criteria within 6 months.
Number of subjects with clinically relevant non-major bleeding events | 0-6 months after randomization
  Number of subjects with clinically relevant non-major bleeding events according to International Society on Thrombosis and Haemostasis criteria within 6 months.
Number of subjects with new intracranial haemorrhage or worsening of the previous intracranial haemorrhage | 0-6 months after randomization
Number of subjects with any bleeding events within 6 months | 0-6 months after randomization

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital Capital Medical University, Beijing, China